CLINICAL TRIAL: NCT05938127
Title: The Impact of Inspiratory Muscle Strength Training and Personalized Exercise Prescription on Metabolism, Cardiovascular Function, and Cardiorespiratory Fitness in Lymphoma Survivors
Brief Title: Impact of Respiratory Training in Lymphoma Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-1216.cc; NCI-2023-03997 (Other: CTRP)
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hodgkin Lymphoma; Non Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Lymphoma Survivors IMST (Experimental): Participants will undergo a version of the BfitBwell Cancer Exercise Program physical assessment, which assesses physical fitness and function.
  Interventions: Device: Inspiratory muscle strength training
- Lymphoma Survivors sham IMST (Experimental): Participants will undergo a version of the BfitBwell Cancer Exercise Program physical assessment, which assesses physical fitness and function.
  Interventions: Device: Sham Inspiratory muscle strength training

INTERVENTIONS:
Device: Inspiratory muscle strength training — High-resistance inspiratory muscle strength training (IMST) is a time-efficient (~5 minutes/day) form of exercise that employs an affordable, handheld device which impedes inspiratory breathing to train the diaphragm and accessory respiratory muscles
  Other Names: IMST
  Arms: Lymphoma Survivors IMST
Device: Sham Inspiratory muscle strength training — Low-resistance inspiratory muscle strength training
  Other Names: Sham IMST
  Arms: Lymphoma Survivors sham IMST

SUMMARY:
High-resistance inspiratory muscle strength training (IMST) is a time-efficient (~5 minutes/day) form of exercise that employs an affordable, handheld device which impedes inspiratory breathing to train the diaphragm and accessory respiratory muscles and has demonstrated improvements in both cardiovascular health (9 mmHg reduction in systolic blood pressure, 45% improvement in vascular endothelial function) and improve exercise tolerance (12% increase in treadmill exercise time) in generally healthy midlife/older adults. Therefore, this approach may circumvent preventative hurdles to exercise, and augment the effects of exercise for capable survivors.

DETAILED DESCRIPTION:
Cancer survivorship has been steadily improving as a result of earlier detection and improved therapies. Behind cancer recurrence, the primary cause of morbidity and mortality among survivors stems from the onset of cardiovascular disease that arises in part due to cardiotoxic chemo and radiation therapies. The increased risk of cardiovascular disease is particularly high in specific survivor populations, such as lymphoma survivors. Although exercise has been demonstrated to improve both recovery after cancer therapy and quality of life, both physical and logistical hurdles may prohibit certain patients from accessing this intervention. High-resistance inspiratory muscle strength training (IMST) is a time-efficient (~5 minutes/day) form of exercise that employs an affordable, handheld device which impedes inspiratory breathing to train the diaphragm and accessory respiratory muscles and has demonstrated improvements in both cardiovascular health (9 mmHg reduction in systolic blood pressure, 45% improvement in vascular endothelial function) and improve exercise tolerance (12% increase in treadmill exercise time) in generally healthy midlife/older adults. Therefore, this approach may circumvent preventative hurdles to exercise, and augment the effects of exercise for capable survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80
* Primary cancer diagnosis of lymphoma
* Able and willing to participate in a supervised exercise program at the Anschutz Health and Wellness Center
* Provides a signed physician exercise clearance form
* SBP > 120 mmHg
* Completion of curative cancer treatment over 12 months prior (individuals on maintenance therapy will be included)
* Possession of a smartphone compatible with the IMST training application (available on both Android and Apple).

Exclusion Criteria:

* oSecond active cancer diagnosis
* oPlanned active cancer treatment or change in current treatment in the next 6 months

  * Severe obesity (BMI >; 40 kg/m2) or underweight (BMI <18.5 kg/m2)
  * Unstable weight (>; 3 kg change in body mass in last 3 months)
  * Significant metabolic disorder (e.g. diabetes type II)
  * Uncontrolled thyroid disease
  * Recent changes in hypertensive medication (within last 3 months)
  * Any medical condition that would impact the safety of, or participation in, an exercise program, including:
  * Significant pulmonary conditions such as chronic obstructive pulmonary disease, emphysema, or interstitial lung disease
  * Known cardiovascular disease, significant hypertension (>180/120), or a recent cardiac event (within past 6 months)
  * Orthopedic conditions such as advanced osteoarthritis, mobility-limiting amputations or chronic injuries, or mobility-limiting acute orthopedic injuries
  * Advanced rheumatoid arthritis or chronic widespread pain conditions such as fibromyalgia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Total Participants Recruited | 2 years
  Count of number of participants recruited into the study
Enrolled Participants per Month | 2 years
  Average number of participants enrolled per month of the study
Valid Assessments per Participant | 5 months
  Adherence to 75% of the program will be deemed acceptable
Session Attendance per Participant | 5 months
  Adherence to 75% of the program will be deemed acceptable
Total Participants Completing the Intervention | 2 years
  Adherence to 75% of the program will be deemed acceptable
Systolic Blood Pressure | 5 months
  Resting systolic blood pressure, collected in triplicate

SECONDARY OUTCOMES:
Molecular Markers - Acetylcholine-stimulated production of nitric oxide | 5 months
  Serum will be used to perform experiments in which purchased cultured endothelial cells will be exposed to 10% serum from human subjects for 24 hours. The investigators will measure acetylcholine-stimulated production of nitric oxide (NO) in endothelial cells following serum incubation. Serum will be collected via venipuncture performed at the CTRC and stored at -80°C until analysis.
Molecular Markers - Acetylcholine-stimulated basal reactive oxygen species production | 5 months
  Serum will be used to perform experiments in which purchased cultured endothelial cells will be exposed to 10% serum from human subjects for 24 hours. The investigators will measure acetylcholine-stimulated basal reactive oxygen species (ROS) production in endothelial cells following serum incubation. Serum will be collected via venipuncture performed at the CTRC and stored at -80°C until analysis.
Cardiorespiratory Fitness (CRF) will be assessed via estimated VO2max | 5 months
  This will be measured by the Tecumseh Step Test. Participants step on and off an 8" step for 3 min, at a metronome-controlled pace of 24 steps/min. Afterward, they immediately sit down, and heart rate is recorded at 30 s and 1 min after completion (using Polar F4 heart rate monitors). These recovery heart rates are then entered into a predictive formula, along with patient biometric information (age, weight, gender), to calculate an estimated VO2max.
Physical function primarily assessed by the 6MWT | 5 months
  Participants will be instructed to walk as far as possible in a six minute period on an indoor track.
Metabolomics analyses will be performed on blood samples | 5 months
  Metabolomics analyses will be performed on blood samples collected during a standardized aerobic exercise session. Samples will be collected before exercise, immediately after, and after 30 min of recovery. Samples will be collected with patient-centric Tasso+ devices (Tasso, Inc) which minimize the discomfort of collection.
Functional Assessment of Cancer Therapy - General (FACT-G, assessing quality of life) | 5 months
  A 27-item scale commonly used to assess overall quality of life in the general cancer survivor population. Scores range from 0-108 with higher scores indicate higher quality of life.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) | 5 months
  A 13-item scale commonly used to assess cancer-related fatigue in cancer survivors. Scores range from 0-52 with higher scores indicate lower levels of fatigue.
Godin Leisure Time Physical Activity Questionnaire | 5 months
  A 6-item scale asking participants the amount of time spent in light, moderate, and vigorous physical activity during the past week. Scores start at 0 with no upper range. Higher scores indicate more minutes of activity per week.
Hospital Anxiety and Depression Scale (HADS) | 5 months
  14 item scale indicating levels of anxiety and depression in clinical populations. Scores range from 0-21 for anxiety and depression scales. Higher scores indicate higher levels of anxiety and depression.
Cardiac risk factors will be collected from medical history forms | 5 months
  These risk factors will be included in secondary analyses to assess if participants at higher known risk of cardiac disease differ in their response to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Marker, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Anschutz Health and Wellness, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No